CLINICAL TRIAL: NCT07063537
Title: Evaluation of the Accuracy and Reproducibility of Visual Field Testing Using a Virtual Reality Head-Mounted Device for Patients With Early, Moderate, and Advanced Glaucoma
Brief Title: Feasibility, Accuracy, and Reproducibility of Virtual Reality Visual Field Testing in Patients With Glaucoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Brennan Eadie, MD, PhD, FRCSC. Assistant Professor, Glaucoma Division; Department of Ophthalmology and Visual Sciences. Dalhousie University, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1030608
Record Dates: First submitted 2025-06-20; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Glaucoma Open-Angle
Keywords: Virtual Reality; Visual Field; Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Intervention Model Description: All participants will perform both a Humphrey visual field test and a virtual reality based visual field test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Visual Field Testing (Experimental): Participants will perform both a virtual reality-based visual field test and a standard Humphrey visual field test for both eyes.
  Interventions: Device: Virtual Reality Visual Field (VR-VF)

INTERVENTIONS:
Device: Virtual Reality Visual Field (VR-VF) — Both devices administer a standard visual field test. The Humphrey is the gold standard desk top model and the VR-VF is a virtual reality headset designed to deliver visual field testing

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of using virtual reality based visual field testing to monitor glaucoma in a clinical setting. This will be done through comparison of a virtual reality (VR) based device to the current gold standard Ziess Humphrey Field Analyzer (HFA). The main questions the study aims to answer are:

* Can both devices produce similar results in terms of detecting visual field defects and progression?
* Does the stage (early, moderate, advanced) of glaucoma impact results between the two devices?

Participants will perform both a standard and a VR based visual field test at each visit, for a total of 5 visits.

DETAILED DESCRIPTION:
The proposed study aims to evaluate the global and pointwise accuracy and reproducibility of a virtual reality (VR) based visual field testing system on a Pico VR platform in direct comparison to the current standard Zeiss Humphrey Field Analyzer (HFA) in glaucoma patients with various levels of decreased visual field sensitivities. Specifically, we aim to evaluate (1) if both devices produce similar global and pointwise threshold values; (2) the reproducibility of threshold values across the entire tested visual field; (3) whether the stage of glaucoma impacts the accuracy and reproducibility between the two devices; (4) whether scotomas exhibit similar threshold sensitives and reproducibility between the two devices; and (5) differences in reported reliability indices between the two devices.

Each participant will perform visual field testing for both eyes using both the VR visual field system and HFA (order randomized). Five separate sessions (both tests for each patient; both eyes) will be conducted, at least 24 hours apart. Patients will also be asked to fill out a questionnaire to qualitatively evaluate their perception of each visual field test.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* diagnosis of primary open-angle glaucoma
* ability to perform visual field testing
* capacity to provide informed consent to research protocol

Exclusion Criteria:

* diagnosis of secondary glaucoma or non-glaucomatous optic neuropathy
* previous intraocular surgery (excluding cataract surgery and minimally invasive glaucoma surgery)
* significant media opacity
* pregnancy
* seizure disorder
* cardiac pacemaker/other implantable device
* severe vertigo/balance disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-14 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Visual field point-wise threshold values | Measured during each visual field test on visits 1 through 5 (throughout study completion, average 2 months)
  Both the VR visual field and HFA produce threshold light sensitivity values measured in decibels (db) at the same locations in space (e.g., 24-2 protocol with stimuli 6 degrees apart at locations up to 30 degrees from central fixation)
Global indices of visual field loss | Measured during each visual field test on visits 1 through 5 (throughout study completion, average 2 months)
  Mean deviation (MD) and pattern standard deviation (PSD) are measurements of global field loss produced by both devices.
Reliability Indices | Measured during each visual field test on visits 1 through 5 (throughout study completion, average 2 months)
  Fixation losses, false positives, false negatives are recorded during each visual field test and reflect the reliability of the given test.

SECONDARY OUTCOMES:
Reliability over time | Measured during each visual field test on visits 1 through 5 (throughout study completion, average 2 months)
  Assessed through examination of variation in global indices and point-wise threshold values
Patient satisfaction | Questionnaire completed at the end of each testing session, following the completion of both visual field tests (throughout study enrolment, average 2 months)
  Patient experience questionnaires will assess the perceived difficulty of performing the test (very difficult, somewhat difficult, neither difficult nor easy, somewhat easy, or very easy), patient comfort during the test (very uncomfortable, somewhat uncomfortable, neutral, somewhat comfortable, or very comfortable), and patient preference between the two devices (conventional visual field test, VR visual field test, or no preference)

CONTACTS AND LOCATIONS:
Overall Officials: Brennan Eadie, MD, PhD, FRCSC, Principal Investigator — Nova Scotia Health
Locations (1):
- Eadie Technologies Inc, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canadian Ophthalmological Society Glaucoma Clinical Practice Guideline Expert Committee; Canadian Ophthalmological Society. Canadian Ophthalmological Society evidence-based clinical practice guidelines for the management of glaucoma in the adult eye. Can J Ophthalmol. 2009;44 Suppl 1:S7-93. doi: 10.3129/cjo44s1. No abstract available. English, French. PMID 19492005
- [Background] Selvan K, Mina M, Abdelmeguid H, Gulsha M, Vincent A, Sarhan A. Virtual reality headsets for perimetry testing: a systematic review. Eye (Lond). 2024 Apr;38(6):1041-1064. doi: 10.1038/s41433-023-02843-y. Epub 2023 Nov 30. PMID 38036608
- [Background] Glen FC, Baker H, Crabb DP. A qualitative investigation into patients' views on visual field testing for glaucoma monitoring. BMJ Open. 2014 Jan 10;4(1):e003996. doi: 10.1136/bmjopen-2013-003996. PMID 24413347
- [Background] Tham YC, Li X, Wong TY, Quigley HA, Aung T, Cheng CY. Global prevalence of glaucoma and projections of glaucoma burden through 2040: a systematic review and meta-analysis. Ophthalmology. 2014 Nov;121(11):2081-90. doi: 10.1016/j.ophtha.2014.05.013. Epub 2014 Jun 26. PMID 24974815